CLINICAL TRIAL: NCT05803824
Title: Efficacy of Baduanjin Qigong Exercise Program on Fatigue and Postural Imbalance Following Lower Limb Burn Injury
Brief Title: Qigong Exercise on Fatigue and Postural Imbalance in Lower Limb Burn Injury
Acronym: Burn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khadra Mohamed Ali, Doctor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2451981
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-03

CONDITIONS: Lower Limb Burn Injury

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A: Baduanjin Qigong exercise plus selected exercise (Experimental): Baduanjin exercise 3 times each week, 30- 60 minutes each time for 12 weeks. The whole set of Baduanjin exercise consists of 9 postures: (1) ready position, (2) holding the hands high with palms up. (3) posing like an archer shooting on left and right sides, (4) holding one arm aloft . (5) looking backwards to prevent sickness and strain, (6) swinging the head and lowering the body t. (7) moving the hands down the back and legs and touching the feet . (8) thrusting the fists and making the eyes glare . and (9) raising and lowering the heels .
  Puls Selected Exercise Program
  * balance exercises is composed of three phases, including warm-up, balance training and cool down.
  * Resisted Exercises were given according to the standardized Oxford technique of progressive resistance exercises .
  Interventions: Other: exercise therapy program
- Patients at group B: patients will receive selected exercise program (Experimental): Selected Exercise Program: Patients will receive
  * balance exercises is composed of three phases, including warm-up, balance training and cool down.
  * Resisted Exercises were given according to the standardized Oxford technique of progressive resistance exercises .
  Interventions: Other: exercise therapy program

INTERVENTIONS:
Other: exercise therapy program — patients will receive Baduanjin Qigong exercise plus selected exercise. the subjects will recive Baduanjin exercise 3 times each week, 30- 60 minutes each time for 12 weeks.
  The whole set of Baduanjin exercise consists of 9 postures: (1) ready position, (2) holding the hands high with palms up. (3) posing like an archer shooting on left and right sides, (4) holding one arm aloft . (5) looking backwards to prevent sickness and strain, (6) swinging the head and lowering the body t. (7) moving the hands down the back and legs and touching the feet . (8) thrusting the fists and making the eyes glare . and (9) raising and lowering the heels .
  Selected Exercise Program: Patients will receive
  * balance exercises is composed of three phases, including warm-up, balance training and cool down.
  * Resisted Exercises were given according to the standardized Oxford technique of progressive resistance exercises

SUMMARY:
90 patients who suffer from chronic fatigue syndrome and postural imbalance following Lower Limb Burn Injury. will be selected from outpatient clinic, faculty of physical therapy, Cairo university. Patients will be assigned randomly into 3 groups of equal numbers, group A: (Study group A) will receive Baduanjin Qigong exercise plus selected exercise program. group B:(Study group B) will receive Baduanjin Qigong exercise, Group C (control group C) will receive selected exercise program .

DETAILED DESCRIPTION:
Patients at group A: patients will receive Baduanjin Qigong exercise plus selected exercise. the subjects practiced Baduanjin exercise 3 times or above each week, 30- 60 minutes each time for 8 weeks. The subjects were required to complete the program in the fixed site and in a collective manner, with special personnel recording the attendance and providing guidance. The whole set of Baduanjin exercise consists of 9 postures: (1) ready position, (2) holding the hands high with palms up to regulate the internal organs, (3) posing like an archer shooting on left and right sides, (4) holding one arm aloft to regulate the functions of the spleen and stomach, (5) looking backwards to prevent sickness and strain, (6) swinging the head and lowering the body to relieve stress, (7) moving the hands down the back and legs and touching the feet to strengthen the kidneys, (8) thrusting the fists and making the eyes glare to enhance strength, and (9) raising and lowering the heels to cure diseases .

Selected Exercise Program: Patients will receive

* balance exercises 3 sessions a week for 8 weeks in the form of balance exercises and resisted exercises. Balance Exercises Each session of balance exercises is composed of three phases, including warm-up, balance training and cool down. The warm-up phase involved gentle stretching for calf, hamstring, quadriceps, iliopsoas muscles, as well as anterior, posterior and lateral step-ups for 5-10 minutes. The active phase was performed on a balance training mat of high-elasticity for 20 minutes. It included heel and toe raises, one-legged stance for each extremity, shifting weight anteriorly, posteriorly, laterally and diagonally. turning head to the right and then to the left with maintaining the feet together, walking in slow motion, step-ups, narrow walking, backward walking, sideward walking, stepping over obstacles, passing balls arranged on the training mat in a circle, and throwing and catching a ball on the training mat. The program ended with 5-10 minutes of cool down. During the cool-down phase, patients performed deep breathing exercises and static exercises for back extensor in a recumbent position.
* Resisted Exercises were given according to the standardized Oxford technique of progressive resistance exercises for hip flexors and extensor, knee extensors and flexors, and ankle dorsiflexors. The exercises' intensity was progressed as the following; week one: 50-60% of three repetition maximum (3RM), from 2nd -6th weeks: 70- 75% of 3RM and for 7th -8th weeks: 80-85% 3RM for 4- 10 repetitions ,3 sessions a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1) age of the patient was ranged from 35 to 55 years; 2) weight range 60-85 kg, height 155- 170 cm; 3) total burned surface area (TBSA) was 20- 35% measured by the rule of nines; 4) the burn cause was thermal; 5) burn depth, partial-thickness burn injury; 6) at least 3 months after burn injuries; 7) and with low physical activity level

Exclusion Criteria:

* 1)inhalation injury; 2) leg amputation; 3) any limitation in LL range of motion; 4) auditory or visual problems; 5) congenital musculoskeletal deformities, especially in the foot; 6) psychiatric disorders; 7) paralysis; or 8) cardiac abnormalities or cardiac pacemakers.

In order to apply the inclusion and exclusion criteria, all cases will be subjected to an interview and assessment.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
The Brief Fatigue Inventory (BFI) | 3months
  The instrument is used to quickly assess the severity of fatigue experienced by cancer patients, as well as its impact on their ability to function over the previous 24 h.he BFI is a reliable and valid tool with a low respondent burden, suitable for measuring fatigue in burn patients during the first year of recovery.
b. The dynamic balance score | 3 months
  c. The dynamic balance score that was measured by the Biodex Balance System (Biodex Medical System, Shirley, NY, USA). Biodex Balance System is a valid and reliable method to assess the dynamic balance. The system has a movable circular platform that permits about 20◦ tilt in 360◦ range so it is free to move about the anterior-posterior and mediallateral directions simultaneously

SECONDARY OUTCOMES:
b. The timed up and go (TUG) test | 3 months
  e. The timed up and go (TUG) test is a basic mobility assessment tool that records the time taken (in seconds) to get up from a chair, walk 3-meter distance, come back and sit down again on the chair
c. The Activities-specific Balance (ABC) scale | 3months
  d. The Activities-specific Balance (ABC) scale is a popular and subjective questionnaire to assess balance confidence and the risk of fall in people with balance problems.34 The ABC scale consisted of 16 items with a total score between 0% (not confident) to 100% (completely confident), where higher scores equate to higher balance confidence and vice versa. The Arabic version of the ABC scale is reliable and valid in the assessment of balance confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan, Principal Investigator — Cairo University
Locations (1):
- faculty of physical therapy , Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
after 6months we will share the study protocol and informed consent.
Supporting Information: Study Protocol, ICF
Time Frame: after 6 months of study